CLINICAL TRIAL: NCT03405909
Title: Standardized Contrast-enhanced Ultrasound (CEUS) -Algorithms for the Non-invasive Diagnosis of Hepatocellular Carcinoma (HCC) in High-risk-patients - a Prospective German Multicenter Study
Brief Title: Standardized CEUS Algorithms for Diagnosis of HCC - Prospective German Multicenter Study
Acronym: ESCULAP
Status: Completed | Type: Observational
Sponsor: University Hospital Erlangen (Other)
Responsible Party: Principal Investigator, Dr. med. Barbara Schellhaas and Prof. Dr. med. Deike Strobel, MD, University Hospital Erlangen
Other Study IDs: DEGUM CEUS HCC
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Hepatocellular Carcinoma; Cholangiocarcinoma, Intrahepatic; Liver Cirrhosis; Liver Cancer; Liver Neoplasms; Liver Diseases
Keywords: contrast-enhanced ultrasound; non-invasive diagnosis; focal liver lesion; liver cirrhosis; standardised diagnostic algorithm; intrahepatic cholangiocellular carcinoma; ESCULAP; CEUS LI-RADS; imaging; hepatocellular carcinoma; MRI; diagnostic accuracy; interobserver agreement; Erlanger Synopsis of CEUS for Liver lesion Assessment in Patients at risk; CEUS Liver Imaging Reporting and Data System
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma; Liver Cirrhosis; Liver Neoplasms; Liver Diseases | interventions — Shadowing Technique, Histology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients at risk for HCC: Patients with any of the following conditions:
  liver cirrhosis of any origin chronic hepatitis B infection chronic hepatitis C infection with advanced fibrosis non-alcoholic steatohepatitis (NASH) hemochromatosis
  Interventions: B-mode ultrasound, contrast enhanced ultrasound (CEUS); MRI / histology
  Interventions: Diagnostic Test: contrast enhanced ultrasound (CEUS); Diagnostic Test: MRI; Diagnostic Test: Histology

INTERVENTIONS:
Diagnostic Test: contrast enhanced ultrasound (CEUS) — CEUS with SonoVue following standardized protocol
Diagnostic Test: MRI — CE-MRI following standardized protocol
Diagnostic Test: Histology — diagnostic liver biopsy

SUMMARY:
Aim of this prospective national multicenter study is to improve standardization of contrast-enhanced ultrasound (CEUS) in the non-invasive diagnosis of hepatocellular carcinoma (HCC) in high-risk patients.

The study is funded by the German Society for Ultrasound in Medicine (DEGUM).

DETAILED DESCRIPTION:
To date, CEUS criteria for non-invasive diagnosis of HCC include arterial phase hyperenhancement, followed by contrast washout in the portal venous or late phase. We would like to investigate the following points:

1. whether arterial hyperenhancement alone is sufficient for the definite diagnosis of HCC in cirrhosis with CEUS
2. whether a further clearly-defined point of assessment in the late phase after 4-6 minutes is of additional diagnostic value in focal liver lesions showing no contrast washout after 3 minutes
3. diagnostic value of CEUS-based standardised diagnostic algorithms (ESCULAP = Erlanger Synopsis of Contrast Enhanced Ultrasound for Liver lesion Assessment in Patients at risk; CEUS LI-RADS = Contrast Enhanced Ultrasound Liver Imaging Reporting and Data System) for non-invasive diagnosis of HCC in high-risk patients (diagnostic accuracy, interobserver-variability, feasability in clinical Routine).

ELIGIBILITY:
Inclusion Criteria:

* high risk for HCC
* focal liver lesion on B-mode ultrasound

Exclusion Criteria:

* pre-treated HCC lesion
* systemic therapy for HCC (sorafenib, regorafenib and others)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High-risk patients for HCC according to German national guidelines (AWMF / DGVS): 1- cirrhosis of any origin; 2- chronic hepatitis B infection; 3 - chronic hepatitis C infection; 4 - non-alcoholic steatohepatitis (NASH); 5 - hereditary hemochromatosis
Sampling Method: Probability Sample
Enrollment: 517 (Actual)
Dates: Start 2018-04-21 (Actual); Primary Completion 2019-04-06 (Actual); Study Completion 2019-04-06 (Actual)

PRIMARY OUTCOMES:
Diagnostic value of standardised CEUS-based algorithms for the non-invasive diagnosis of HCC in high-risk patients | 2 years
  Diagnostic accuracy, interobserver-variabilty and feasability in clinical routine for CEUS-based algorithms Reference Standard: histology / MRI

SECONDARY OUTCOMES:
Diagnostic value / dispensability of contrast washout for definite diagnosis of HCC with CEUS | 2 years
  Sensitvity, specificity, positive and negative predictive value of arterial hyperenhancement only compared with arterial hyperenhancement followed by contrast washout for non-invasive diagnosis of HCC in high-risk patients Reference Standard: histology / MRI
Standardisation of CEUS examinations | 2 years
  Diagnostic value of an additional standardised examination point in the late phase after 4-6 minutes in lesions without contrast washout after 3 minutes Reference Standard: histology / MRI
Diagnostic accuracy of CEUS in intrahepatic cholangiocellular carcinoma (ICC) | 2 years
  Sensitvity, specificity, positive and negative predictive value of contrast-enhanced ultrasound for non-invasive diagnosis of ICC in high-risk patients / differential diagnosis of HCC versus ICC Reference Standard: histology
Comparison of two CEUS-based algorithms | 2 years
  ESCULAP versus CEUS LI-RADS (diagnostic accuracy, interobserver agreement) Reference Standard: histology / MRI
Non-inferiority of CEUS versus MRI for non-invasive diagnosis of HCC | 2 years
  Comparison of CEUS and MRI for non-invasive diagnosis of HCC (diagnostic accuracy, interobserver agreement) Reference Standard: histology
Influence of histological grading on contrast enhancement behaviour | 2 years
  correlation of histological grading and contrast enhancement pattern

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Schellhaas, MD, Principal Investigator — University Hospital Erlangen, Department of Medicine 1; Deike Strobel, MD, Principal Investigator — University Hospital Erlangen, Department of Medicine 1
Locations (1):
- University Hospital Erlangen, Department of Medicine 1, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No